CLINICAL TRIAL: NCT02797769
Title: Risk of Cardiovascular Events in Patients Using Tocilizumab as Compared With Other Biologics in Multiple Large Healthcare Databases
Brief Title: A Time to Cardiovascular Event Analysis Comparing Tocilizumab to Other Biologics in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: GA30048
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Non-TNFi Biologics: Real world patients with RA with a dispensing history for non-TNFi biologics (such as abatacept or tofacitinib) will be included.
  Interventions: Drug: Other Biologics
- TNFi Biologics: Real world patients with RA with a dispensing history for TNFi biologics will be included.
  Interventions: Drug: Other Biologics
- Tocilizumab: Real world patients with RA with a dispensing history for tocilizumab will be included.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Other Biologics — Exposure data will be gathered from claims databases, and no medicine will be administered in this non-interventional study. There are no protocol-specified biologic agents, although the analyses will be stratified by TNFi and non-TNFi targeted therapies. The drug selection and regimen are at the discretion of the prescribing physician.
  Groups: Non-TNFi Biologics; TNFi Biologics
Drug: Tocilizumab — Tocilizumab exposure data will be gathered from claims databases, and no medicine will be administered in this non-interventional study. The regimen is at the discretion of the prescribing physician.
  Other Names: Actemra
  Groups: Tocilizumab

SUMMARY:
This retrospective cohort study will analyze data from multiple large U.S. health insurance claims databases to compare use of tocilizumab to other biologic disease-modifying anti-rheumatic drugs (DMARDs) in real world patients with RA. Using the date of dispensing as the index date, the analysis will compute the time to first event for several cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 inpatient or 2 outpatient diagnoses of RA
* Continuous medical/pharmacy coverage and full claims data available
* At least 6 months of insurance plan enrollment prior to index date

Exclusion Criteria:

* Nursing home residents
* Human immunodeficiency virus (HIV)
* Malignancy
* Receipt of chemotherapy
* End-stage renal disease, dialysis, or transplant
* Use of rituximab
* Recent cardiovascular event (includes MI, stroke, ACS, or HF) within 90 days prior to index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real world patients with RA who received tocilizumab or other biologic therapy will be included. Data will be collected from multiple large U.S. health insurance claims databases in this retrospective cohort analysis.
Sampling Method: Non-Probability Sample
Enrollment: 48950 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
Time to First Event of Myocardial Infarction (MI) or Stroke with Tocilizumab Versus Tumor Necrosis Factor Inhibitor (TNFi) Therapies | Up to approximately 1 year from index date

SECONDARY OUTCOMES:
Time to First Event of MI or Stroke with Tocilizumab Versus Non-TNFi Therapies | Up to approximately 1 year from index date
Time to Hospitalization for Coronary Revascularization Procedure | Up to approximately 1 year from index date
Time to Hospitalization for Acute Coronary Syndrome (ACS) | Up to approximately 1 year from index date
Time to First Event of MI, Stroke, Coronary Revascularization Procedure, or ACS | Up to approximately 1 year from index date
Time to Heart Failure (HF) Requiring Hospitalization | Up to approximately 1 year from index date
Time to All-Cause Death | Up to approximately 1 year from index date

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

REFERENCES:
- [Result] Kim SC, Solomon DH, Rogers JR, Gale S, Klearman M, Sarsour K, Schneeweiss S. No difference in cardiovascular risk of tocilizumab versus abatacept for rheumatoid arthritis: A multi-database cohort study. Semin Arthritis Rheum. 2018 Dec;48(3):399-405. doi: 10.1016/j.semarthrit.2018.03.012. Epub 2018 Mar 22. PMID 29673963
- [Result] Kim SC, Solomon DH, Rogers JR, Gale S, Klearman M, Sarsour K, Schneeweiss S. Cardiovascular Safety of Tocilizumab Versus Tumor Necrosis Factor Inhibitors in Patients With Rheumatoid Arthritis: A Multi-Database Cohort Study. Arthritis Rheumatol. 2017 Jun;69(6):1154-1164. doi: 10.1002/art.40084. Epub 2017 Apr 28. PMID 28245350